CLINICAL TRIAL: NCT00542230
Title: High Sensitivity Screening of Compound Libraries to Discover a Drug for the Treatment of Sickle Cell Disease
Brief Title: Blood Sampling for Research Related to Sickle Cell Disease
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080004; 08-DK-0004
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-10-27

CONDITIONS: Sickle Cell Trait; Sickle Cell Disease; Sickle Cell Anemia
Keywords: Erythrocytes; Drug Screen; Sickle Cell Trait; Sickle Hemoglobin; Sickle Cell Disease; Natural History
MeSH Terms: conditions — Sickle Cell Trait; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Healthy Volunteers
- Sickle Cell Trait: Patient with sickle cell trait or disease

SUMMARY:
This study will collect representative blood samples from healthy children and adults and from children and adults who have unique red blood cell features that are related to sickle cell disease. Sickle cell disease is a blood disease that limits the ability of red blood cells to carry oxygen throughout the body. The purpose of the study is to collect a variety of blood samples that may then be used to investigate advances and potential new drug treatments for sickle cell disease.

Volunteers must be at least 18 years of old. Samples will be taken both from healthy volunteers and from volunteers who have unique red blood cell features that are related to sickle cell disease. Candidates will be screened with a medical history.

During the study, participants will undergo a one- to two-hour outpatient procedure at the National Institutes of Health Clinical Center. Once researchers have explained the study and obtained the participant s consent, participants will donate 8 cc (approximately 2 teaspoons) of blood.

Because repeat testing helps researchers validate study findings, participants who have the unique red blood cell features mentioned above may also be asked if they are willing to return and donate another 2 cc to 8 cc of blood for additional studies. The amount of blood drawn will not exceed 50 ml with any eight-week period for adults or 7 cc within any six-week period for children.

DETAILED DESCRIPTION:
The critical event leading to serious morbidity in sickle cell disease is polymerization of the abnormal hemoglobin to form fibers that stiffen and distort red blood cells and consequently, cause vaso-occlusion in the small vessels of the tissues. Currently, hydroxyurea is the only approved drug for treating sickle cell disease, but is only partially effective. This protocol seeks to identify by high sensitivity in vitro screening methods additional compounds that inhibit sickling. Subjects with sickle cell trait or disease and normal volunteers will be asked to donate blood samples for studies to verify their hemoglobinopathies and then periodically donate small volume samples of fresh blood for use in ongoing high throughput screening tests to identify potentially clinically useful anti-sickling drugs.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with sickle cell trait
* Patients with known hemoglobinopathies involving one or two genes for sickle hemoglobin
* Healthy volunteers for control experiments
* Age range: adults greater than or equal to 18 years of age

EXCLUSION CRITERIA:

* Subjects who are unable to comprehend the investigational nature of the laboratory research are ineligible to enroll in this protocol.
* As a safety precaution in handling the blood samples, patients with HIV, Hepatitis B or Hepatitis C will be excluded from the study. HIV, Hepatitis B or Hepatitits C testing will not be done under this study. Participants must be co-enrolled under another NIH protocol where the screening evaluation has been performed.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2007-11-07 (Actual)

PRIMARY OUTCOMES:
To screen large compound libraries for anti-sickling activity, particularly compounds that are already FDA-approved drugs, with the goal of discovering a drug for treating sickle cell disease. | daily
  To identify by high sensitivity in vitro screening methods additional compounds that inhibit sickling

CONTACTS AND LOCATIONS:
Overall Officials: William A Eaton, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2008-DK-0004.html